CLINICAL TRIAL: NCT00005708
Title: Improving Adherence to Interventions for Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4917; R01HL051119 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To develop effective strategies for enhancing adherence to therapeutic interventions designed to improve care for hypertensive minority populations.

DETAILED DESCRIPTION:
BACKGROUND:

The study was in response to a demonstration and education initiative, "Improving Hypertensive Care for Inner City Minorities", which was reviewed and approved by the Clinical Applications and Prevention Advisory Committee in April 1992 and by the National Heart, Lung, and Blood Advisory Council in May 1992. The Request for Applications was released in October 1992.

DESIGN NARRATIVE:

An aggressive Hypertension Intervention Project (HIP) was developed in the Hypertension Research Section of King/Drew Medical Center in South-Central Los Angeles. The private CHUER clinic (located in the same cachement area) subcontracted with the Drew University Center in a community coalition consisting of several large health advocacy organizations. All subjects were randomized into usual care (controls) or interventional care (experimental) at the initiation of the HIP. The cornerstone of the aggressive intervention was the development of a computerized patient tracking system and the introduction into the clinic of several educational activities including a) exit interviews; b) home visits; c) support group sessions, and d) community health seminars/fairs. Community Health Workers performed the bulk of the patient tracking and educational intervention field work. Outcome measures of pre and post-study blood pressure, renal function, body weight change, and all-cause mortality were compared between experimental and controls at two, three and four years into the study. Quality-of-life questionnaires were obtained pre- and post-study and analyzed for new insights into needs assessment, awareness of hypertension, attitudes towards treatment, compliance with drug therapy, and effectiveness of various educational interventions employed in the study. Concurrent efforts to reduce co-morbid risk factors such as obesity, cigarette smoking, excessive alcohol consumption and stress were assessed as secondary outcomes. The HIP hoped to demonstrate cost-effective innovations for the adaptation of these Medical Center-targeted strategies to community physicians and health clinics of the inner city.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1997-08 (Actual)

REFERENCES:
- [Background] Ward HJ, Morisky DE, Lees NB, Fong R. A clinic and community-based approach to hypertension control for an underserved minority population: design and methods. Am J Hypertens. 2000 Feb;13(2):177-83. doi: 10.1016/s0895-7061(99)00149-1. PMID 10701818